CLINICAL TRIAL: NCT02971579
Title: A Network on the Quality of ERCP, on the Organization of the Endoscopic Units and on the Training of the Endoscopists in Italy
Brief Title: A Register on the Quality of ERCP and Training of Endoscopists in Italy
Acronym: REQUEST
Status: Completed | Type: Observational
Sponsor: ASST Rhodense (Other)
Responsible Party: Principal Investigator, gianpiero manes, MD, ASST Rhodense
Other Study IDs: request
Record Dates: First submitted 2016-11-20; First posted 2016-11-23 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Biliary Tract Diseases; Pancreatic Diseases
Keywords: ERCP; biliary diseases; Pancreatic diseases; outcome; Quality; Training
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases; Gallbladder Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ERCP — Endoscopic procedure used to manage biliary and pancreatic diseases

SUMMARY:
This is a prospective observational longitudinal study

Aim of the study is to collect information:

* on the organization models of the Endoscopic Units performing ERCP in Italy
* on the previous and/or ongoing training of the endoscopists performing ERCP
* on the clinical characteristics of patients undergoing ERCP in Italy as well as on the outcome

DETAILED DESCRIPTION:
Quality of ERCP in Italy has been object of various, mainly retrospective studies in Italy, but it has never systematically and prospectively evaluated in a large prospective series.

Moreover, the study aim at collecting data on the organization models of the Endoscopic Units performing ERCP in Italy; on the previous and/or ongoing training of the endoscopists performing ERCP; on the clinical characteristics of patients undergoing ERCP in Italy as well as on the outcome of the procedure

The study consists of 3 phases:

1. Collection of the information on the Endoscopic Unit and on the endoscopists who performed ERCP in the center
2. Collection of data regarding consecutive ERCPs performed in adult patients in each center including demographic, clinical and procedural information
3. Definition of the the outcome of ERCP assessed after 30 days from the procedure

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study

Exclusion Criteria:

* Informed consent not subscribed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing ERCP for various indications
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Complications rate | 30 days
  Occurrence of post -ERCP complications

SECONDARY OUTCOMES:
Rate of repeated procedure | 30 days
  The rate of ERCPs that have to be repeated within 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Occhipinti, MD, Principal Investigator — AOU Maggiore della Carità Novara
Locations (1):
- AOU Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No